CLINICAL TRIAL: NCT00844324
Title: A Single Dose, 2-Period, Cross-over, Bioequivalence Study in Healthy Subjects to Evaluate the Proposed Commercial Oral Suspension of Candesartan Cilexetil
Brief Title: Bioequivalence Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: James Hainer, Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D2451C00007
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension
Keywords: Candesartan; Bioequivalence
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Candesartan cilexetil 1mg/mL
  Interventions: Drug: Candesartan cilexetil
- B (Experimental): Candesartan cilexetil 1.6mg/mL
  Interventions: Drug: Candesartan cilexetil

INTERVENTIONS:
Drug: Candesartan cilexetil — Formulation:Oral suspensionStrength:1 mg/mLDose: 32 mg, single dose
  Arms: A
Drug: Candesartan cilexetil — Formulation:Oral suspensionStrength:1.6 mg/mLDose: 32 mg, single dose
  Arms: B

SUMMARY:
This study is designed as a Phase-I, 2-period, cross-over, randomised, open-label, single centre study to determine bioequivalence of a single 32 mg dose of the proposed commercial oral suspension of candesartan cilexetil (1 mg/mL) and a single 32 mg dose of the candesartan cilexetil oral suspension (1.6 mg/mL) used in the paediatric program.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Body mass index (BMI) 19-27 kg/m2 calculated from height and weight at the Screening visit
* Clinically normal physical findings including ECG and safety laboratory values at the Screening visit and on Day -1 of each treatment period, including negative results for drugs-of-abuse, alcohol, Hepatitis B, Hepatitis C and HIV.

Exclusion Criteria:

* History of significant mental, cardiac, renal, hepatic or significant gastrointestinal disease (that may affect the rate and extent of absorption of the IP), as judged by the Investigator
* Any condition which could modify the absorption of the IPs
* Previous randomisation of treatment in the present study
* History or symptoms and signs of ongoing severe allergic disease/hypersensitivity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
PK (Candesartan cilexetil) | Collected at pre-dose and at selected time points; 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 30 and 36 hours post-dose

SECONDARY OUTCOMES:
Safety variables (adverse events, ECG, vital signs, safety laboratory) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: James Hainer, MD, Study Director — AstraZeneca; Klaus Francke, Dr, Principal Investigator — Parexel
Locations (1):
- Research Site, Harrow, United Kingdom